CLINICAL TRIAL: NCT00199303
Title: Efficacy of Pre- and Post-Operative Oral Dextromethorphan for Reduction of Intra- and 24-Hr Post-Operative Morphine Consumption for Transabdominal Hysterectomy
Brief Title: Efficacy of Pre- and Post-Operative Oral Dextromethorphan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: efficacy of dextromethorphan; KhonKaen University
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2002-07

CONDITIONS: Efficacy of Dextromethorphan; Morphine Consumption; Pain
Keywords: NMDAreceptor antagonist, dextromethorphan; pain, post-operative; opioid consumption, morphine
MeSH Terms: conditions — Pain; Pain, Postoperative

INTERVENTIONS:
Drug: pre-operatively followed by 30 mg three times per day after surgery

SUMMARY:
We studied the effect of dextromethorphan (DEX), an N-methyl-d-aspartate antagonist, on analgesic consumption and pain scoring after abdominal hysterectomy. Our aim was to compare the analgesic effectiveness and incidence of adverse side effects of oral DEX with placebo (P)

DETAILED DESCRIPTION:
One hundred patients were randomized to two groups. Group DEX was given 30 mg tablets of oral dextromethorphan with their pre-medication and three more times in the first 24 hours after surgery. Group P received the placebo following the same schedule. Post-operative analgesic requirements were assessed using a patient-controlled analgesia system.

Pain was assessed at rest using a visual analog scale in the post anesthetic care unit(PACU), 6 and 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 30 and 60, with an ASA physical status of I or II, undergoing elective total abdominal hysterectomy under general anesthesia.

Exclusion Criteria:

* Women with a history of significant renal or hepatic impairment, allergy to any of the study medications, antitussive or NSAID use (48 hours or 1 week, respectively) before surgery, chronic pain and regular analgesic use, were excluded. Patients taking medications that could interact with dextromethorphan, including quinidine, flecainide, mexiletine, fluoxetine, amitriptyline, nortriptyline, and propafenone

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2002-12; Study Completion 2003-12

PRIMARY OUTCOMES:
Mean morphine consumption
Mean pain score

CONTACTS AND LOCATIONS:
Overall Officials: waraporn chau-in, Asso Prof., Study Chair — Department of Anesthesiology, Faculty of Medicine,KhonKaen University,KhonKaen 40002, Thailand; BUSABONG SUKMOUEN, Dr., Principal Investigator — Department of Anesthesiology; KRIANGSAK NGAMSANGSIRISAPT, Dr., Principal Investigator — Department of Anesthesiology; WINITA JIRARAREUNGSAK, Principal Investigator — Department of Anesthesiology
Locations (1):
- Waraporn Chau-in, KhonKaen, KhonKaen, Thailand